CLINICAL TRIAL: NCT05272046
Title: Comparison of the Performance of Monopolar Current Cutting Knife and Bipolar RFA Knife in POEM (Per-Oral Endoscopic Myotomy)
Brief Title: Monopolar and Bipolar Current RFA Knife in POEM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Salmaan Azam Jawaid, MD, Principal Investigator, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H-50587
Record Dates: First submitted 2022-02-04; First posted 2022-03-09 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Esophageal Motility Disorders
Keywords: Achalasia; Dysphagia; Per-Oral Endoscopic Myotomy; Bipolar electrocautery
MeSH Terms: conditions — Esophageal Motility Disorders; Esophageal Achalasia; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Two groups with patients randomized into receiving either the standard of care bipolar electrocautery tool or monopolar electrocautery tool.
Who Masked: Participant
Masking Description: Patient will not know which electrocautery tool will be used in their procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Monopolar Electrocautery tool (Active Comparator): Patients randomized into this group will receive the standard of care monopolar tool for their POEM procedure.
  Interventions: Procedure: Per-oral Endoscopic Myotomy
- Bipolar Electrocautery tool (Experimental): Patients randomized into this group will receive the standard of care bipolar tool for their POEM procedure.
  Interventions: Procedure: Per-oral Endoscopic Myotomy; Device: Speedboat (Bipolar electrocautery knife)

INTERVENTIONS:
Procedure: Per-oral Endoscopic Myotomy — Therapeutic endoscopy procedure by means of electrocautery surgical tools for treatment of various esophageal conditions such as achalasia or spastic esophageal disorders.
  Other Names: POEM
Device: Speedboat (Bipolar electrocautery knife) — Use of Creo Medical's Speedboat RS2 knife and generator in performing the POEM procedure for patients presenting with an esophageal motility disorder.
  Other Names: Speedboat Inject
  Arms: Bipolar Electrocautery tool

SUMMARY:
Per Oral Endoscopic Myotomy (POEM) is performed for various esophageal muscular disorders, including achalasia and other spastic esophageal conditions. It is performed with the standard endoscope and involves dissecting the esophageal muscle sphincter. The procedure is typically completed using standard monopolar energy, which are effective, but can be associated with post-procedural pain. More importantly, frequent exchange of various instruments are required in order to cut the right layers and to stop bleeding. The Speedboat-RSD is FDA approved for dissection of various tissue within the gastrointestinal tract tract but only a few studies have evaluated its use in POEM. Currently, the investigators have been performing EGD with POEM procedures using Speedboat-RSD as a standard of care procedure. The investigators would like to compare the performance of the standard monopolar ERBE knife to the bipolar Speedboat-RSD knife in POEM. The investigators hypothesize the bipolar knife will allow for efficient completion of the POEM procedure with less post procedural pain.

DETAILED DESCRIPTION:
Per Oral Endoscopic Myotomy (POEM) is performed for various esophageal motility disorders, including achalasia and other spastic esophageal conditions. It is performed with the standard endoscope and involves dissection of the esophageal submucosa followed by cutting of the esophageal muscle. The procedure is typically completed using standard monopolar cutting knives, which are effective, but can be associated with inadvertent thermal injury and post-procedural pain due to dissemination of higher voltage. More importantly, frequent exchange of various instruments are required in order to inject within the submucosa and to coagulate bleeding vessels. The Speedboat-RSD has an integrated injection needle for submucosal injection and uses bipolar radiofrequency energy (BRF) and microwave energy to dissect tissue/coagulate vessels. In essence, injection, submucosal dissection, cutting, and coagulation can all occur with one knife (2). It is FDA approved for submucosal dissection (ESD) and myotomy within the gastrointestinal tract but only a few studies have evaluated its use in POEM (3). Currently, the investigators have been performing EGD with the POEM procedure using Speedboat-RSD as a standard of care procedure. The investigators would like to compare the performance of the standard monopolar ERBE knife to the bipolar Speedboat-RSD knife in POEM. The investigators hypothesize the bipolar knife will allow for efficient completion of the POEM procedure with less post-procedural related pain.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years of age
* Able to sign consent - Planned POEM procedure for all indications

Exclusion Criteria:

* Pregnant patients
* Prisoners
* Unable to sign consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2025-02-19 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain score | Pre-procedure, 1-hour post procedure, 8-10 hours post procedure, and 24 hours post procedure.
  Use of a Visual Analog Scale (VAS) from 0-10 with "0" being no pain and "10" being the worse pain to assess overall pain following the POEM procedure up to 24 hours.

SECONDARY OUTCOMES:
Technical success rate of patients who completed POEM procedure with the bipolar knife. | Day 1
  Completion of POEM procedure with the Speedboat-RS2 knife
Total procedure time (minutes) | Day 1
  Includes time from incision, tunneling, dissection and closure.
Study knife removal during procedure | Day 1
  Total number of times the Speedboat knife needed to be removed for another device during mucosal incision, submucosal dissection, or myotomy.
Hospital Length-of-stay | Up to 1 week
  Number of days patient remains in hospital following procedure
Adverse events | 1 month, 3 months, 6 months, and 12 months.
  Collection of unanticipated medical occurrences within a 12 month time frame.

CONTACTS AND LOCATIONS:
Locations (3):
- Baylor College of Medicine, Houston, Texas, United States
- Asian Institute of Gastroenterology (AIG) Hospitals, Hyderabad, India
- Navarra Hospital Complex - Navarra Hospital, Pamplona, Spain

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.

REFERENCES:
- [Background] Jung D, Youn YH, Jahng J, Kim JH, Park H. Risk of electrocoagulation syndrome after endoscopic submucosal dissection in the colon and rectum. Endoscopy. 2013 Sep;45(9):714-7. doi: 10.1055/s-0033-1344555. Epub 2013 Aug 29. PMID 23990482
- [Background] Saunders B P, Tsiamoulos Z P, Bourikas L et al.The
- [Background] Patil G, Dalal A, Maydeo AP. Feasibility of Speedboat RS2 with bipolar radiofrequency energy for peroral endoscopic myotomy in patients with achalasia (with video). Endosc Int Open. 2020 Aug;8(8):E998-E1001. doi: 10.1055/a-1165-0087. Epub 2020 Jul 21. PMID 32743048